CLINICAL TRIAL: NCT07399327
Title: Biomarkers of Response to SEEG Thermocoagulation in Patients With Refractory Focal Epilepsy
Brief Title: Biomarkers of Response to SEEG Thermocoagulation
Acronym: THALPO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: CRMBM-CEMEREM (Unknown); UMR 5203, InsermU1191, IGF, Montpellier (Unknown); Aix Marseille Université (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RCAPHM24_0270; ID-RCB 2025-A00344-45 (Other: ANSM)
Record Dates: First submitted 2026-01-06; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Drug Resistant Epilepsy
Keywords: RFTC; Drug resistant epilepsy; SEEG
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Patient Health Questionnaire; myotrophin; Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SEEG patients (Experimental)
  Interventions: Other: Quality of life questionnaires (QOLIE, EFIQUACEE for children), psychiatric questionnaires (NDDIE, GAD-7, PCL-5) at Visit 1 (V1), V5, V6 and V7; Other: Resting state SEEG recording 30min before and 30 min after RFTC; Other: Blood sample at Visit 1 (V1), V2, V4 and V5; Other: SEEG electrodes tissue-traces sample at V3 (during SEEG electrodes ablation); Other: Multiparametric 3T MRI with gadolinium at V1, V4 and V5; Other: Multiparametric 7T MRI at V1 and V5

INTERVENTIONS:
Other: Quality of life questionnaires (QOLIE, EFIQUACEE for children), psychiatric questionnaires (NDDIE, GAD-7, PCL-5) at Visit 1 (V1), V5, V6 and V7 — This intervention consists in the completion of diverse questionnaires assessing the quality of life of the subject. These questionnaires include:
  * quality of life questionnaires: QOLIE or EFICACEE for children
  * psychiatric questionnaires NDDIE, GAD-7, PCL-5 These questionnaires will be performed during V1, V5, V6 and V7
Other: Resting state SEEG recording 30min before and 30 min after RFTC — During this intervention a resting state SEEG recording will be performed before and after RFTC. These recordings will last for 30 minutes each.
Other: Blood sample at Visit 1 (V1), V2, V4 and V5 — Blood samples will be collected at Visit 1 (V1), V2, V4 and V5. 2 tubes of 2 ml EDTA will be collected during these visits
Other: SEEG electrodes tissue-traces sample at V3 (during SEEG electrodes ablation) — During this intervention, investigators will collect brain tissue samples on SEEG electrodes during their extraction.
Other: Multiparametric 3T MRI with gadolinium at V1, V4 and V5 — 3T MRI with gadolinium injections will be performed at V1, V4 and V5.
Other: Multiparametric 7T MRI at V1 and V5 — Patients will undergo 7T MRI at V1 and V5

SUMMARY:
Drug-resistant focal epilepsy is a severe neurological disease that affects one-third of patients with epilepsy. Surgery is the only potentially curative treatment. Intracerebral exploration by stereo electroencephalography (SEEG) is an important step in the surgical pathway. It aims to establish the precise mapping of the epileptogenic network (EZN), including all the brain regions that generate seizures. At the end of SEEG, SEEG-guided radiofrequency thermocoagulation (SEEG RFTC) represents a therapeutic option that may be efficient as a palliative treatment in patients ineligible for resective surgery, or may lead, in some cases, to a definitive effect, avoiding open surgery. The safety and effectiveness of this approach have been established. However, the odds of remaining seizure-free after one year vary greatly between studies, ranging from 4% to 71%. This disparity in therapeutic responses could be linked to the absence of objective criteria for the selection of targets, but also to the existence of mechanisms of action outside of the direct lesional effect. A decrease in SEEG markers of epileptogenicity may predict thermocoagulation efficiency. However, no data are available regarding changes in alteration of the blood-brain barrier (BBB) connectivity, inflammation, or associated molecular changes and their relationship to prognosis.

This study aims to elucidate the mechanisms underlying the clinical effect of SEEG RFTC by studying the changes in electrophysiological (SEEG), structural (ultra-high field MRI), and biological (blood biomarkers of neuro-glio-vascular damage and inflammation, molecular adaptations) markers. They will be correlated with clinical outcome in a prospective cohort of patients with drug-resistant focal epilepsy. As advantages for clinical care, this study will allow selection of RFTC targets based on scientifically validated criteria, and elaboration of predictive scores for therapeutic response in each patient.

The primary objective is to study the predictive factors of response to SEEG RFTC, by correlating changes in BBB permeability with clinical response 3 months after RFTC, in a prospective cohort of patients with drug-resistant focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient, parents or legal representative who have given their written informed consent,
* Adult or pediatric patient ≥ 12 years old suffering from drug-resistant focal epilepsy,
* Standardized pre-surgical assessment including medical history, scalp video-EEG and 3T MRI,
* Patients in whom a SEEG exploration for pre-surgical evaluation has been indicated,
* Patient able to understand, speak and write in French,
* Patient able to follow study's procedure,
* Patient beneficiary or affiliated to a health insurance plan.

Exclusion Criteria:

* Epilepsy surgery performed without the requirement of SEEG,
* Contraindication to 3T or 7T brain MRI (patient with a cardiac pacemaker, metallic foreign bodies, non-removable implanted electronic medical devices, claustrophobia, inability to remain in supine position, patient havingwith Vagus Nerve Stimulation (VNS) or Deep Brain Sstimulation (DBS), intrauterine devices or tattoos in the imaging area less than 6 weeks old at the time of the 3T/7T brain MRI),
* Contraindication to gadolinium-based MRI contrast agent (history of allergic or anaphylactic reaction to gadolinium, hypersensitivity to gadoteric acid, meglumine, or any drug containing gadolinium, severe renal failure (glomerular filtration rate, GFR, below 30 ml/min/1.73 m2), patients on dialysis or with a history of kidney disease, such as renal transplantation, a single kidney, or renal malignancy),
* Person protected by articles L1121-5, L1121-6 and L1121-8 of the Public Health Code (pregnant or breastfeeding woman, deprived of liberty by judicial decision, situations of social fragility, adults unable or unable to express their consent),
* Patient in exclusion period of another study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between changes in the MRI biomarker of BBB permeability (the transfer coefficient, Ki) and clinical response (responder vs non responder) at 3 months after RFTC | From baseline before SEEG to 3 months after RFTC
  Correlation between changes in the MRI biomarker of BBB permeability (the transfer coefficient, Ki), assessed using 3T MRI before SEEG and 3 months after RFTC and clinical response (responder, non-responder) at 3 months after RFTC.

SECONDARY OUTCOMES:
Relationship between changes in MRI biomarkers of microstructural damage, large-scale 7T structural connectivity and functional connectivity response at 3 months after RFTC. | From baseline before SEEG to 3 months after RFTC.
  Correlation between changes in MRI biomarkers of microstructural damage (7T T1 longitudinal relaxation time, T2* effective transversal relaxation time, and tissue susceptibility), large-scale 7T structural connectivity (connectivity strengths assessed using DWI MRI) and functional connectivity (Pearson's correlation coefficient using BOLD resting state fMRI) assessed using 7T MRI before SEEG and 3 months after RFTC, and the clinical response (responder, non responder) at 3 months after RFTC.
Relationship between changes in MRI biomarkers of BBB permeability, microstructural damage, large-scale 7T structural connectivity and functional connectivity and clinical response at 6-12 months after RFTC. | From baseline before SEEG to 6 months and 12 months after RFTC
  Correlation between changes in MRI biomarkers of BBB permeability (transfer coefficient, Ki), microstructural damage (7T T1 longitudinal relaxation time, T2* effective transversal relaxation time, and tissue susceptibility), structural connectivity (connectivity strengths assessed using DWI MRI), functional connectivity (Pearson's correlation coefficient using BOLD resting state fMRI), assessed using 3T/7T MRI before SEEG and 3 months after RFTC, and the clinical response (responder vs. non responder; percentage change in seizure frequency) at 6 months and 12 months after RFTC
Relationship between changes in interictal SEEG-biomarkers (spikes- and HFO rates, power spectrum density (PSD), functional connectivity and clinical response at 3, 6 and 12 months after RFTC. | From 30 minutes before to 30 minutes after RFTC for SEEG biomarkers; from baseline before SEEG to 3, 6 and 12 months after RFTC for clinical response.
  Correlations between changes in interictal SEEG-biomarkers (spikes and HFO rates, power spectrum density (PSD), functional connectivity assessed by non-linear correlation coefficient h2) after RFTC versus before RFTC and clinical response (responder vs non responder; percentage change in seizure frequency versus baseline before SEEG) at 3, 6 and 12 months after RFTC.
Relationship between changes in blood biomarkers within 72h and 3 months after RFTC and clinical response at 3, 6 and 12 months after RFTC. | From baseline to 72 hours and 3 months after RFTC for blood biomarkers; from baseline to 3, 6 and 12 months after RFTC (radiofrequency thermocoagulation) for clinical response
  Correlation between changes in blood biomarkers (including GFAP, S100b, NFL, UHCL1) within 72 hours and 3 months after RFTC versus before SEEG and clinical response (responder vs non responder; percentage change in seizure frequency versus baseline before SEEG) at 3, 6 and 12 months after RFTC.
Changes in epileptogenicity markers within and outside the Epileptogenic Zone Network (EZN) 24 hours after RFTC | Within 24 hours after RFTC (during SEEG electrode ablation)
  Comparison of omic profiles, specifically ictal epileptogenicity markers EI (Epileptogenicity Index) cEI (connectivity Epileptogenicity Index) and PEI (Permutation Entropy Index) within and outside the Epileptogenic Zone Network (EZN) 24 hours after RFTC
Changes from baseline in the quality of life questionnaire scores at 3-6-12 months after RFTC. | From baseline before SEEG to 3 months, 6 months and 12 months after RFTC.
  Changes in QOLIE scale (Quality of Life in Epilepsy Inventory-Form 31, 0 to 100, 100 being the best outcome) for adults or EFIQUACCE (its equivalent for children) from baseline, which were assessed before SEEG and at 3, 6, and 12 months after RFTC.
To compare between groups the psychiatric impact (depression and anxiety) | From baseline before SEEG to 3 months, 6 months and 12 months after RFTC
  Changes between groups of psychiatric comorbidities, specifically depression: score of the NDDI-E (Neurological Disorders Depression Inventory for Epilepsy, 6 to 24, 24 meaning bad outcome), PCL-5 (Post-Traumatic Stress Disorder Checklist for DSM-5, 0 to 52, 52 being the worst outcome) and anxiety: Score of GAD-7 (Generalized Anxiety Disorder - 7, between 0 and 21, 21 meaning bad outcome)

IPD SHARING:
Plan to Share IPD: No